CLINICAL TRIAL: NCT02799186
Title: PREVALENCE STUDY OF FIBROMUSCULAR DYSPLASIA IN PATIENTS WITH HAEMATOMA OR SPONTANEOUS CORONARY ARTERY DISSECTION
Brief Title: The Study of the Prevalence Fibromuscular Dysplasia in Patient With Haematoma or Spontaneous Coronary Artery Dissection.
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Heart and Research Foundation (Unknown); French Coronary Atheroma and Interventional Cardiology Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0267; 2016-A00403-48 (Registry Identifier: 2016-A00403-48)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2016-06

CONDITIONS: Spontaneous Coronary Artery Dissection; Spontaneous Coronary Artery Haematoma
Keywords: Spontaneous Coronary Artery Dissection; haematoma; Fibromuscular Dysplasia; genetic analysis; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Hematoma; Fibromuscular Dysplasia; Acute Coronary Syndrome | interventions — Blood Specimen Collection; Genetic Testing

ARMS (1):
- SCAD (spontaneous coronary artery dissection) (Experimental): Every patient included with a SCAD or hematoma, will systematic benefit a tomographic or MRI angiography of renal, cerebrovascular and iliac arteries, to look for the presence of a fibromuscular displasia. A blood sample will be collected for the genetic analysis which will be realized by the Team 3 of the INSERM UMR970, Paris Cardiovascular research Center, France.
  Interventions: Procedure: blood sample for genetic analysis

INTERVENTIONS:
Procedure: blood sample for genetic analysis

SUMMARY:
Spontaneous Coronary Artery Dissection (SCAD) is a rare and often misdiagnosed cause of Acute Coronary Syndrome (ACS) affecting predominantly young women without cardiovascular risk factors. The origin of SCAD remains uncertain but a strong and frequent association with Fibromuscular Dysplasia (FMD) has been recently reported based on imaging evidence only.

The aim of our study is to assess the presence of FMD and its genetic determinants i in a sample for haematoma or spontaneous coronary artery dissection.

From May 2016 to 2018 we plan to include prospectively and retrospectively 200 patients admitted for ACS with confirmed diagnosis of SCAD. This study will be conducted in more than 30 French interventional cardiology centers. Coronary angiograms or intracoronary imaging data will be reviewed by two experienced interventional cardiologist experts in SCAD diagnosis.

For each patient a genetic analysis will be performed. A systematic screening for FMD will be realized by computed tomographic or MRI angiography of renal, cerebrovascular and iliac arteries and reviewed by two experienced radiologists. A one year follow-up is expected.

This study aims to confirm the presumed association of FMD and SCAD through the exploration of several artery beds and the study of confirmed genetic determinants, which has never been described previously to our knowledge.

DETAILED DESCRIPTION:
The recruitment of patients takes place in each interventional cardiology department.

The patients can be included in a retrospective way (for SCAD occurred from 2010) or forward-looking way. The patients are informed about this study by the investigator. After a reflection period and an answer to the possible questions, the patient is included. The informed consent is signed.

Every patient included with a SCAD or hematoma, will systematic benefit a tomographic or MRI angiography of renal, cerebrovascular and iliac arteries, to look for the presence of a fibromuscular displasia. A blood sample will be collected for the genetic analysis which will be realized by the Team 3 of the INSERM UMR970, Paris Cardiovascular research Center, France.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria :

* Patients over 18 year's old
* Patient with a possible diagnosis of spontaneous coronary dissection defined by:

  * A picture of SCA
  * Compatible angiographic signs
  * More or less confirmed by intracoronary imaging (OCT/IVUS) or check angiographic control (upper to 1 month)
* Patient having given his informed consent and signed to participate to the study
* Subject accepting the use of its personal data in the form of an anonymous codification including in the scientific publications.

Exclusion Criteria:

* - Minor patient
* Major patient submitted to a protective measure (guardianship, supervision guardianship)
* No affiliation to the French social security system
* Coronary dissection with traumatic or iatrogenic origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of the SCAD in the population of patients taken care for a ACS | at day 1

SECONDARY OUTCOMES:
Prevalence of the FMD in the population SCAD from a tomographic or MRI angiography analysis of renal, cerebrovascular and iliac arteries | at day 1
Hormonal Parameters ( gynecological factors) | at day 1
Environmental Factors : physical exercise or an recent intense emotional stress | at day 1
Genetic Factors (including recently identified genetic risk loci for FMD) | at day 1
Morbi-mortality to 1 year | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pascal MOTREFF, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France